CLINICAL TRIAL: NCT03529409
Title: Hybrid Effectiveness-Implementation Trial for ART Adherence and Substance Use in HIV Care in South Africa
Brief Title: Effectiveness & Implementation of a Behavioral Intervention for Adherence and Substance Use in HIV Care in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Cape Town (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jessica Magidson, Assistant Professor, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187/2018; K23DA041901 (NIH)
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Results first posted 2021-10-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Human Immunodeficiency Virus; Alcohol-Related Disorders; Drug Use
Keywords: Immunologic Deficiency Syndromes; Substance Use; Acquired Immunodeficiency Syndrome; Immune System Diseases; Behavioral Symptoms; RNA Virus Infections; HIV Infections; Alcohol Use; Drug Use
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol-Related Disorders; Immunologic Deficiency Syndromes; Substance-Related Disorders; Immune System Diseases; Behavioral Symptoms; RNA Virus Infections; HIV Infections; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project Khanya (Experimental): Those assigned to Project Khanya (the behavioral intervention for substance use and adherence condition) will have approximately 6 sessions (including Life-Steps, behavioral activation, and relapse prevention) delivered by a peer interventionist plus standard of care, which is typically referral to a local outpatient substance use treatment clinic. They will also receive a Wisepill, a wireless, real-time adherence monitoring device.
  Interventions: Behavioral: Project Khanya
- ESOC (No Intervention): Those assigned to the ESOC (enhanced standard of care) condition will receive the standard of care, which is referral to a local substance use treatment clinic. The substance use clinics in the location that this study occurs follow the Matrix, and evidence-based 16-week outpatient program to treat substance use. We will enhance patients' normal referral to Matrix for ESOC participants by promoting facilitating and following up on the referral. Additionally, those in the control group will also receive a Wisepill, a wireless adherence monitoring device.

INTERVENTIONS:
Behavioral: Project Khanya — This treatment involves integrating a behavioral intervention for substance use with a behavioral intervention for adherence.
  Arms: Project Khanya

SUMMARY:
The purpose of this study is to test the effectiveness and implementation of a brief, integrated behavioral intervention for HIV medication adherence and substance use in the HIV care setting in South Africa. The intervention is specifically designed to be implemented by non-specialist counselors using a task sharing model in local HIV clinics. The behavioral intervention will be compared to usual care, enhanced with referral to a local outpatient substance use treatment program (Enhanced Standard of Care - ESOC) on study endpoints (as described in study endpoint section below).

DETAILED DESCRIPTION:
The HIV epidemic in South Africa (SA) is among the highest in the world. SA has a large antiretroviral therapy (ART) program, but some individuals exhibit poor ART adherence, which increases the likelihood of developing drug resistance and failing the only available first and second line ART regimens in SA. ART nonadherence contributes to greater morbidity, mortality, and higher likelihood of sexual HIV transmission when virus is detectable. At the same time, alcohol and other drug use is prevalent among HIV-infected individuals in SA and associated with worse ART adherence, lower rates of viral suppression, and HIV transmission risk behavior. Yet, despite the impact of untreated substance use on poor HIV treatment outcomes and continued HIV transmission, there is little if any integration of substance use and HIV care services in SA, which creates a fragmented and incomplete system of care. This study had three phases, first being formative, qualitative work which led to a systematic treatment adaptation phase. This third phase, the clinical trial, is based on this formative work and other empirical support using behavioral interventions to improve ART adherence and reduce substance use in resource-limited settings, including SA. This study is a Type 1 hybrid effectiveness-implementation trial of a lay counselor-delivered behavioral intervention for adherence and substance use integrated into the HIV primary care setting in SA. To ensure that those who need this intervention most will receive it, participants will be patients with HIV who are struggling with adherence (as defined in the investigator's inclusion criteria) and who have an elevated substance use risk.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive and on ART
* 18-65 years of age
* Elevated substance use risk (ASSIST score greater than or equal to 4 for drugs or greater than or equal to 11 for alcohol)
* Have at least one of the following:

  1. Not attained viral suppression from first line ART (VL>400 copies/mL)
  2. On second-line ART treatment
  3. Reinitiated first-line treatment within the past three months
  4. Had a pharmacy non-refill at least once in the past 3 months

Exclusion Criteria:

* Inability to provide informed consent or complete procedures in English or isiXhosa
* Severe risk/likely dependence for opiates (ASSIST score >26) because opiate substitution therapy may not be available
* Severe alcohol dependence symptoms that may warrant medical management of potential withdrawal symptoms
* Active, untreated, major mental illness (with untreated psychosis or mania) that would interfere with the paraprofessional adapted intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica F Magidson, PhD, Principal Investigator — University of Maryland
Locations (2):
- University of Maryland, College Park, Maryland, United States
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses are complete, de-identified data will be available per request of outside individual.

REFERENCES:
- [Derived] Lu T, Belus JM, Majokweni S, Joska J, Regenauer KS, Rose AL, Myers B, Burnham W, Andersen LS, Ryan DA, Cadet T, Magidson JF, Murphy SM. Cost-effectiveness of a peer-delivered behavioral intervention for adherence to antiretroviral therapy and alcohol and drug use in South African HIV care. AIDS Care. 2026 Jan 22:1-10. doi: 10.1080/09540121.2026.2613989. Online ahead of print. PMID 41567004
- [Derived] Belus JM, Anvari MS, Ke H, Regenauer KS, Ma T, Myers B, Andersen LS, Joska JA, Magidson JF. Effects of HIV and alcohol stigma on biomarker-confirmed alcohol use following a peer-delivered intervention in South Africa. Addict Behav Rep. 2025 Nov 1;22:100640. doi: 10.1016/j.abrep.2025.100640. eCollection 2025 Dec. PMID 41312191
- [Derived] Belus JM, Regenauer KS, Lu T, Murphy SM, Rose AL, Ochieng YA, Joska J, Majokweni S, Andersen LS, Myers B, Safren SA, Magidson JF. Increases in employment over six months following Khanya: A secondary analysis of a pilot randomized controlled trial of a peer-delivered behavioral intervention for substance use and HIV medication adherence in Cape Town, South Africa. Int J Drug Policy. 2024 Dec;134:104632. doi: 10.1016/j.drugpo.2024.104632. Epub 2024 Nov 21. PMID 39577326
- [Derived] Belus JM, Rose AL, Andersen LS, Ciya N, Joska JA, Myers B, Safren SA, Magidson JF. Adapting a Behavioral Intervention for Alcohol Use and HIV Medication Adherence for Lay Counselor Delivery in Cape Town, South Africa: A Case Series. Cogn Behav Pract. 2022 May;29(2):454-467. doi: 10.1016/j.cbpra.2020.10.003. Epub 2020 Nov 10. PMID 36171964
- [Derived] Belus JM, Joska JA, Bronsteyn Y, Rose AL, Andersen LS, Regenauer KS, Myers B, Hahn JA, Orrell C, Safren SA, Magidson JF. Gender Moderates Results of a Randomized Clinical Trial for the Khanya Intervention for Substance Use and ART Adherence in HIV Care in South Africa. AIDS Behav. 2022 Nov;26(11):3630-3641. doi: 10.1007/s10461-022-03765-8. Epub 2022 Jul 27. PMID 35895150
- [Derived] Magidson JF, Joska JA, Belus JM, Andersen LS, Regenauer KS, Rose AL, Myers B, Majokweni S, O'Cleirigh C, Safren SA. Project Khanya: results from a pilot randomized type 1 hybrid effectiveness-implementation trial of a peer-delivered behavioural intervention for ART adherence and substance use in HIV care in South Africa. J Int AIDS Soc. 2021 Jun;24 Suppl 2(Suppl 2):e25720. doi: 10.1002/jia2.25720. PMID 34164935
- [Derived] Magidson JF, Joska JA, Myers B, Belus JM, Regenauer KS, Andersen LS, Majokweni S, O'Cleirigh C, Safren SA. Project Khanya: a randomized, hybrid effectiveness-implementation trial of a peer-delivered behavioral intervention for ART adherence and substance use in Cape Town, South Africa. Implement Sci Commun. 2020;1:23. doi: 10.1186/s43058-020-00004-w. Epub 2020 Mar 4. PMID 32607502

RESULTS

PARTICIPANT FLOW:
Groups:
- Pre-Randomization: Participants enrolled in the study at the baseline assessment, but who were never randomized (approximately 2 weeks post-baseline) and therefore did not continue with the study.
Period: Randomized
Arm/Group | Project Khanya | ESOC | Pre-Randomization
Started | 30 | 31 | 5
Completed | 30 | 31 | 0
Not Completed | 0 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 4
Not completed — Excluded | 0 | 0 | 1
Period: Post-treatment Assessment
Arm/Group | Project Khanya | ESOC | Pre-Randomization
Started | 30 | 31 | 0
Completed | 26 | 26 | 0
Not Completed | 4 | 5 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Unable to contact for this assessment, but attended later assessments | 2 | 4 | 0
Period: Follow-up Assessment
Arm/Group | Project Khanya | ESOC | Pre-Randomization
Started | 28 (All participants were eligible for Follow-Up regardless of Post-Treatment attendance.) | 30 (All participants (n=31) were eligible for Follow-Up regardless of Post-Treatment attendance) | 0
Completed | 27 | 29 | 0
Not Completed | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-Randomization: Participants enrolled in the study at the baseline assessment, but who were never randomized (approximately 2 weeks post-baseline) and did not continue with the study.
- Total: Total of all reporting groups
Arm/Group | Project Khanya | ESOC | Pre-Randomization | Total
Number analyzed (Participants) | 30 | 31 | 5 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.80 (10.47) | 34.29 (7.99) | 31.60 (9.56) | 36.59 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 3 | 36
  Male | 17 | 11 | 2 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black African | 29 | 31 | 5 | 65
  Mixed race | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 30 | 31 | 5 | 66
HIV medication adherence [Mean (Standard Deviation); unit: percentage of days adherent] — Population: HIV medication adherence was assessed between baseline and randomization visits. As the pre-randomization participants did not attend randomization, HIV medication adherence could not be calculated.
  percentage of days adherent
    number analyzed (Participants) | 30 | 31 | 0 | 61
    (all) | 53.6 (32.1) | 49.3 (29.8) |  | 46.60 (31.56)
Positive alcohol or drug urine test result [Count of Participants; unit: Participants] | 27 | 29 | 4 | 60
Phosphatidylethanol (PEth) concentration [Mean (Standard Deviation); unit: ng/ML] — Objective biomarker of alcohol use that can detect blood collected up to 21 days after alcohol consumption. Minimum detection value is 8 ng/mL. Higher PEth values indicate greater concentration of alcohol. Values of ≥ 50 ng/mL indicate unhealthy drinking.
  ng/ML | 686.0 (639.9) | 456.1 (530.8) | 370.8 (418.4) | 554.1 (582.0)
Moderate or high-risk on Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) measure [Count of Participants; unit: Participants] — World Health Organization measure used to assess substance use risk for alcohol, cannabis, cocaine, opiates, and amphetamines, hallucinogens, and other drugs. Standardized cutoff scores are used to categorize risk levels: low risk (0-3 for illicit drugs/0-10 for alcohol), moderate risk (4-26 for illicit drugs/11-26 for alcohol), or high risk (> 26) for substance use-related problems.
  Participants | 30 | 31 | 5 | 66
Suppressed viral load, <400 copies/ml [Count of Participants; unit: Participants] | 15 | 24 | 3 | 42
Consumed any substance on timeline followback [Mean (Standard Deviation); unit: percentage of days] | 38.81 (24.58) | 29.49 (21.72) | 42.86 (35.36) | 37.74 (24.29)
Number of drinks on days drinking on timeline followback [Mean (Standard Deviation); unit: number of drinks] — Population: One participant did not complete the measure because reported no alcohol consumption
  number of drinks
    number analyzed (Participants) | 30 | 30 | 5 | 65
    (all) | 7.17 (3.79) | 8.03 (5.59) | 5.37 (6.24) | 7.43 (4.86)

OUTCOME MEASURES:

1. Primary Outcome: Changes in HIV Medication Adherence Throughout Intervention Phase
Description: Percentage of prescribed antiviral therapy agent (medications) taken as measured by real time wireless motoring device
Time Frame: Assessed between baseline assessment and the acute outcome (approximately 12-weeks post-randomization/ post-intervention assessment)
Measure: Mean (Standard Deviation); unit: percentage of days adherent to Wisepill
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 30 | 31
percentage of days adherent to Wisepill | 60.0 (37.1) | 28.2 (32.1)
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .01, Mixed Models Analysis; Mean Difference (Net) = -.287, 95% CI 2-sided [-.507 to -.066]

2. Primary Outcome: Biological Measure of Substance Use
Description: Substance use measured with urinalysis.
Time Frame: Assessed at the acute outcome (approximately 12-weeks post-randomization/ post-intervention assessment)
Measure: Count of Participants; unit: Participants
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 26 | 26
Participants
  Positive | 25 | 23
  Negative | 1 | 3
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .28, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.55. The estimate below is for post-treatment, comparing TAU to Khanya; Mean Difference (Net) = 1.95, 95% CI 2-sided [-1.61 to 5.50]

3. Primary Outcome: Biological Measure of Substance Use
Description: Substance use measured with phosphatidylethanol (PEth) concentration, which is an objective biomarker of alcohol use that can detect blood collected up to 21 days after alcohol consumption. Minimum detection value is 8 ng/mL. Higher PEth values indicate greater concentration of alcohol. Values of ≥ 50 ng/mL indicate unhealthy drinking.
Time Frame: Assessed at the acute outcome (approximately 12-weeks post-randomization/ post-intervention assessment)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 26 | 25
ng/mL | 484.2 (398.7) | 414.7 (389.6)
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .16, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.38. The estimate below is for post-treatment, comparing TAU to Khanya; Mean Difference (Net) = 157, 95% CI 2-sided [-67 to 382]

4. Primary Outcome: Changes in Self-reported Substance Use
Description: World Health Organization Alcohol, Smoking, and Substance Involvement Screening Test (WHO-ASSIST). It is a measure used to assess substance use risk for alcohol, cannabis, cocaine, opiates, and amphetamines, hallucinogens, and other drugs. Standardized cutoff scores are used to categorize risk levels: low risk (0-3 for illicit drugs/0-10 for alcohol), moderate risk (4-26 for illicit drugs/11-26 for alcohol), or high risk (> 26) for substance use-related problems.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 26 | 26
Participants
  moderate or high risk | 23 | 25
  low risk | 3 | 1
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .77, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.90. The estimate below is for post-treatment, comparing TAU to Khanya; Mean Difference (Net) = .25, 95% CI 2-sided [-1.51 to 2.00]

5. Secondary Outcome: Biological Measure of Substance Use
Description: Substance use measured with urinalysis.
Time Frame: Assessed at follow-up (approximately 24-weeks post-randomization/ 6-month follow-up assessment)
Measure: Count of Participants; unit: Participants
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 27 | 29
Participants
  Positive | 20 | 24
  Negative | 7 | 5
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .63, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.55. The estimate below is for follow-up, comparing TAU to Khanya; Mean Difference (Net) = .71, 95% CI 2-sided [-2.24 to 3.67]

6. Secondary Outcome: Biological Measure of Substance Use
Description: as for outcome 3
Time Frame: Assessed at follow-up (approximately 24-weeks post-randomization/ 6-month follow-up assessment)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 25 | 29
ng/mL | 538.4 (554.4) | 386.1 (392.6)
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .44, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.38. The estimate below is for follow-up, comparing TAU to Khanya; Mean Difference (Net) = 84, 95% CI 2-sided [-136 to 304]

7. Secondary Outcome: Changes in Self-reported Substance Use
Description: as for outcome 4
Time Frame: Assessed between baseline assessment and follow-up (approximately 24-weeks post-randomization/ 6-month follow-up assessment)
Measure: Count of Participants; unit: Participants
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 27 | 29
Participants
  moderate or high risk | 24 | 22
  low risk | 3 | 7
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .87, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.90. The estimate below is for follow-up, comparing TAU to Khanya; Mean Difference (Net) = -.16, 95% CI 2-sided [-1.85 to 1.58]

8. Secondary Outcome: Intervention Acceptability
Description: 15-item acceptability subscale of a pragmatic, quantitative assessment based on RE-AIM developed by the Applied Mental Health Research group (AMHR) at Johns Hopkins University. Total scores are averaged across all items and range from 0 to 3. Higher scores indicate greater acceptability.
  Qualitative interviews will also be conducted with intervention participants at the end of the study to assess acceptability guided by RE-AIM and the Proctor model.
Time Frame: Assessed at the acute outcome (approximately 12-weeks post-randomization/ post-intervention assessment)
Measure: Mean (Standard Deviation); unit: average score on a scale
Arm/Group | Project Khanya
Number analyzed (Participants) | 26
average score on a scale | 2.98 (.04)

9. Secondary Outcome: Intervention Feasibility
Description: 14-item feasibility subscale of a pragmatic, quantitative assessment based on RE-AIM developed by the Applied Mental Health Research group (AMHR) at Johns Hopkins University. Total scores are averaged across all items and range from 0 to 3. Higher scores indicate greater feasibility.
  Qualitative interviews will also be conducted with intervention participants at the end of the study to assess feasibility guided by RE-AIM and the Proctor model.
Time Frame: Assessed at the acute outcome (approximately 12-weeks post-randomization/ post-intervention assessment)
Measure: Mean (Standard Deviation); unit: average score on a scale
Arm/Group | Project Khanya
Number analyzed (Participants) | 26
average score on a scale | 2.98 (.18)

10. Secondary Outcome: Intervention Fidelity
Description: Independent fidelity ratings of a randomly selected subset (20%) of intervention sessions using a fidelity assessment developed for each session that includes 15-19 items that map onto each core intervention component, and factors unique to the peer delivery implementation strategy (i.e., appropriate self-disclosure, stigmatizing behaviors, common factors including warmth and non-judgment).
Time Frame: Assessed between randomization and the acute outcome (approximately 12-weeks post-randomization/ post-intervention assessment)
Measure: Mean (Standard Deviation); unit: Percentage fidelity to treatment
Units Other Than Participants: Treatment session recordings
Arm/Group | Project Khanya
Number analyzed (Participants) | 19
Number analyzed (Treatment session recordings) | 36
Percentage fidelity to treatment | 91.7 (13.3)

11. Secondary Outcome: Intervention Uptake
Description: Intervention participant attendance and retention (i.e., the mean number of intervention sessions attended by intervention participants)
Time Frame: as for outcome 10
Measure: Mean (Standard Deviation); unit: Sessions attended
Arm/Group | Project Khanya
Number analyzed (Participants) | 30
Sessions attended | 4.77 (1.96)

12. Other Pre Specified Outcome: HIV Viral Load
Description: Percentage of patients with a suppressed viral load (<400 copies/ml)
Time Frame: Assessed at follow-up (approximately 24-weeks post-randomization/ 6-month follow-up assessment)
Measure: Count of Participants; unit: Participants
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 27 | 29
Participants
  Suppressed | 16 | 22
  Unsuppressed | 11 | 7
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .65, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.89. The estimate below is for follow-up, comparing TAU to Khanya; Mean Difference (Net) = -.47, 95% CI 2-sided [-2.49 to 1.55]

13. Other Pre Specified Outcome: Changes in Self-reported Substance Use
Description: Changes in percent days used any substance measured by timeline follow-back
Time Frame: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of days used any substance
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 27 | 29
percentage of days used any substance | 30.7 (25.9) | 25.1 (23.2)
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .63, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.66. The estimate below is for follow-up, comparing TAU to Khanya; Mean Difference (Net) = 3.3, 95% CI 2-sided [-10.5 to 17.1]

14. Other Pre Specified Outcome: Changes in Self-reported Substance Use
Description: Changes in number of drinks measured by timeline follow-back
Time Frame: as for outcome 7
Measure: Mean (Standard Deviation); unit: number of drinks on days drinking
Arm/Group | Project Khanya | ESOC
Number analyzed (Participants) | 27 | 29
number of drinks on days drinking | 4.61 (3.29) | 4.96 (4.25)
Statistical Analysis 1: Comparison: Project Khanya vs ESOC; Test type: Superiority; p = .85, Mixed Models Analysis — The overall omnibus test of the time by treatment interaction was p=.94. The estimate below is for follow-up, comparing TAU to Khanya; Mean Difference (Net) = -.03, 95% CI 2-sided [-.34 to .28]

ADVERSE EVENTS:
Time Frame: While participants were active in the study (informed consent at baseline assessment until 6-month follow-up; approximately 6 months)
Arm/Group | Project Khanya | ESOC | Pre-Randomization
All-Cause Mortality (participants affected / at risk) | 2/30 | 0/31 | 0/5
Serious Adverse Events (participants affected / at risk) | 8/30 | 0/31 | 1/5
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project Khanya (N=30) | ESOC (N=31) | Pre-Randomization (N=5)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Planned surgery, not study related
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Hospitalization (General disorders) | 1 (2) | 0 (0) | 0 (0) — Hospitalized for cancer diagnosis and treatment
Death (General disorders) | 2 (2) | 0 (0) | 0 (0) — One death due to cancer. One death due to unknown circumstances.
Hospitalization (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hospitalization (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03529409/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03529409/SAP_001.pdf